CLINICAL TRIAL: NCT05744336
Title: Assessing the Impact of Immersive Virtual Reality Experience on Injection-related Anxiety in Patients Undergoing Interventional Pain Spine Procedures: a Prospective Randomized Trial
Brief Title: Impact of Virtual Reality on Anxiety in Patients Undergoing Interventional Procedures
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Jason Ross, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU00218462
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Anxiety
Keywords: Anxiety; Pain Procedures; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled observational trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Immersive Virtual Reality (VR) (Experimental): Participants in Group 1 Immersive Virtual Reality (VR) will wear the device covering their eyes. The viewing experience will include calming nature sounds for between 15-20 minutes before their planned plain clinic procedure.
  Interventions: Other: Group 1 Immersive Virtual Reality (VR)
- Group 2 control group (Placebo Comparator): Group 2 control group has no preprocedural intervention. Standard clinic waiting conditions for 15-20 minutes before their planned pain clinic procedure.
  Interventions: Other: Group 2 Control Group

INTERVENTIONS:
Other: Group 1 Immersive Virtual Reality (VR) — Participants in Group 1 Immersive Virtual Reality (VR) participants wear the device covering their eyes. The viewing experience will include calming nature sounds for between 15-20 minutes before their planned plain clinic procedure
  Arms: Group 1 Immersive Virtual Reality (VR)
Other: Group 2 Control Group — Group 2 control group participants have no preprocedural intervention. Standard clinic waiting conditions for 15-20 minutes before their planned pain clinic procedure.
  Arms: Group 2 control group

SUMMARY:
Periprocedural anxiety is a common problem for patients who undergo interventional pain procedures. Virtual Reality (VR) is an immersive experience that has gained acceptance in the medical field as a tool for reducing anxiety and pain for patients.Research Aim:

To evaluate the effect of immersive virtual reality (VR) on periprocedural anxiety related to therapeutic cervical epidural steroid injections (ESI).

The investigators hypothesize that immersive virtual reality will result in a clinically meaningful anxiety reduction, defined as the proportion of participants with > 50% reduction in Numeric Rating Scale (NRS) anxiety scores when compared to participants in the non-treatment group who will have standard preprocedural waiting time conditions in clinic, but no VR experience. Similarly, the investigators hypothesize a significant reduction in objective sympathetic tone as measured by skin sympathetic nerve activity (SKNA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old at day of enrollment
* Neck pain patient deemed to be a candidate for pain control treatment with interventional fluoroscopically guided cervical epidural steroid injection as determined by their pain medicine provider based on history, physical exam, and radiographic findings
* Willingness to undergo pre-procedural intervention of VR viewing experience or equivalent pre-procedural wait time
* No history of prior epidural steroid injections
* Did not receive sedatives prior to or during procedure

Exclusion Criteria:

* Refusal / inability to participate or provide consent
* Contraindications to injection (anticoagulated states, allergy to components of injection, local infection at injection site, current infectious process or treatment of antibiotics for current infection)
* Uncontrolled anxiety disorder or untreated/inadequately treated psychiatric disorder
* History of Alzheimer's, dementia, or cognitive dysfunction
* Patient currently taking benzodiazepines
* Severe motion sickness
* Seizure disorder
* Vision loss
* Non-English speaking patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric rating score for anxiety while positioning on the fluoroscopy table. | Before planned procedure
  Numeric rating score for anxiety on an 11-point scale, ranging from 0 (no anxiety at all) to 10 (worst possible level of anxiety) when positioning on the fluroscopy table.
Numeric rating score for anxiety when local anesthetic is injected. | Start of planned procedure
  Numeric rating score for anxiety on an 11-point scale, ranging from 0 (no anxiety at all) to 10 (worst possible level of anxiety) when local is injected.
Numeric rating score for anxiety when the epidural needle is removed. | End of planned procedure
  Numeric rating score for anxiety on an 11-point scale, ranging from 0 (no anxiety at all) to 10 (worst possible level of anxiety) after the epidural needle is removed

SECONDARY OUTCOMES:
Procedural pain during epidural steroid injection reported by participants. | During planned procedure
  NRS Level of subjective procedural pain during epidural steroid injection recorded by numeric rating score on a scale of 0 (no pain) to 10 (worst pain imaginable) Level of subjective procedural pain during epidural steroid injection recorded by NRS
Timepoint at peak of numeric rating score anxiety rating | Through study completion average of 2 hours
  Timepoint at peak numeric rating score for anxiety (NRS) 0 (no anxitey) to 10 (worst anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Jason Ross, MD, Principal Investigator — Northwestern Univesity
Locations (1):
- Anesthesiology Pain Medicine Center, Chicago, Illinois, United States